CLINICAL TRIAL: NCT06887205
Title: Immediate Lymphatic Reconstruction After Lymphadenectomy in Melanoma Patients: a Parallel Cohort Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-1357; NCI-2025-01923 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Lymphatic Reconstruction; Lymphadenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper extremity group recieving ALND (Experimental): Participants will be recruited pre-operatively by their treating physicians.
  Interventions: Procedure: Lymphovenous bypass (LVB)
- Lower extremity group getting ILND (Experimental): Participants will be recruited pre-operatively by their treating physicians.
  Interventions: Procedure: Lymphovenous bypass (LVB)

INTERVENTIONS:
Procedure: Lymphovenous bypass (LVB) — At the time of axillary lymph node dissection (ALND) or inguinal lymph node dissection (ILND) in the melanoma patient population.

SUMMARY:
To learn if LBP can help to prevent lymphedema when it is performed at the time of surgery rather than after a patient has already developed the disease.

DETAILED DESCRIPTION:
To examine if performing lymphovenous bypass (LVB) at the time of axillary lymph node dissection (ALND) or inguinal lymph node dissection (ILND) in the melanoma participant population impacts the period prevalence of lymphedema occurrence one year from surgery. To assess wound complications rates occurring in first 30-days post operatively from the time of surgery. To estimate time to drain removal. To estimate the point prevalence of LE following surgery at 3 months, 6 months, and 1 year following surgery. To estimate the cumulative incidence associated with the first appearance of LE. To assess quality of life and survivorship, using Lymphedema Quality of Life (LYMQOL) questionnaire over the study follow-up domain.

ELIGIBILITY:
Inclusion Criteria:

1. Participants greater than or equal to 18 years of age.
2. Participants willing to participate.
3. Participants able to complete informed consent.
4. Participants with a diagnosis of Melanoma undergoing ALND or ILND.

Exclusion Criteria:

1. Participant staking anticoagulants within 7 days prior to surgery.
2. Participants that are known to be pregnant at the time of surgery.
3. Participants with BMI greater than 50.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-09-06 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Ashleigh M Francis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org